CLINICAL TRIAL: NCT02850588
Title: TransCarotid Revascularization Surveillance Project of the Society for Vascular Surgery Vascular Quality Initiative
Brief Title: SVS VQI TransCarotid Revascularization Surveillance Project
Acronym: VQI-TCAR
Status: Recruiting | Type: Observational
Sponsor: Society for Vascular Surgery Patient Safety Organization (Other)
Responsible Party: Sponsor
Other Study IDs: VQI TCAR
Record Dates: First submitted 2016-07-22; First posted 2016-08-01 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Carotid Artery Disease
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TCAR treatment: All patients, both high risk and standard risk surgical patients undergoing transcarotid revascularization with a carotid stent during carotid artery flow reversal in hospitals that participate in the Carotid Artery Stent Registry of the Society for Vascular Surgery Patient Safety Organization
  Interventions: Procedure: Transcarotid artery revascularization
- CEA treatment: All patients undergoing carotid endarterectomy in hospitals that participate in the Carotid Endarterectomy Registry of the Society for Vascular Surgery Patient Safety Organization
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Transcarotid artery revascularization — Direct implantation of a stent into the carotid artery via a surgical incision in the neck combined with blood flow reversal in the carotid artery during stent placement
  Groups: TCAR treatment
Procedure: Carotid endarterectomy — Removal of carotid atherosclerotic plaque (endarterectomy) via a surgical incision in the neck
  Groups: CEA treatment

SUMMARY:
The VQI TCAR Surveillance Project is designed to monitor the safety and effectiveness of stents placed directly into the carotid artery while reversing blood flow within the carotid artery to reduce stroke risk. It will compare this less-invasive surgical procedure with standard carotid endarterectomy in centers that participate in the Society for Vascular Surgery Vascular Quality Initiative.

DETAILED DESCRIPTION:
Background:

Contemporary randomized trials of transfemoral carotid artery stenting (TF CAS) and carotid endarterectomy (CEA) have shown comparable long-term ipsilateral stroke prevention (>30 days) but have consistently demonstrated higher periprocedural (< 30 day) stroke rates, including contralateral stroke, compared with CEA, with the highest risk centered around "day zero". Potential etiologies for this excess risk likely relate to embolization during unprotected catheterization of the aortic arch and supraaortic vessels from a TF approach and/or suboptimal distal embolic protection during CAS. TransCarotid Artery Revascularization (TCAR) combines the surgical principles of neuroprotection with minimally invasive endovascular techniques to treat stenosis in the carotid artery. It involves surgical exposure and clamping of the proximal common carotid artery with continuous carotid blood flow reversal via an extracorporeal arteriovenous shunt from the target carotid artery to a femoral vein, during which carotid bifurcation/internal carotid artery stenting is performed. Thus, TCAR avoids catheter manipulation in the aortic arch and emulates the "clamp and backbleed" method of neuroprotection during CEA, but differs from CEA in that the carotid artery is accessed through a smaller, supra-clavicular incision below the main plexus of cranial nerves. Further, the direct transcarotid approach allows the use of larger bore sheaths and tubing to achieve higher reverse carotid artery flow rates than is possible with smaller transfemoral catheters.

Published TCAR Data:

The initial study of TCAR in patients deemed to be at high risk for complications from CEA have shown that TCAR appears to provide superior stroke and death outcomes when compared to prior registry results from both CEA and TF CAS. Schermerhorn, et al reported outcomes from the Society for Vascular Surgery (SVS) Vascular Registry in high surgical risk patients and found that in this real world registry, the 30-day stroke and death rates in symptomatic patients for CEA and TF CAS were 6.4% and 7.9% respectively. (Citation: Schermerhorn) In asymptomatic, high risk patients, the 30-day stroke and death rates for CEA and TF CAS were 3.7% and 4.8% respectively. In contrast, a recent study of TCAR (ROADSTER pivotal trial) , the 30-day stroke and death rates for both symptomatic and asymptomatic patients were 2.8% and 2.9%, respectively. (Citation: Kwolek) While these initial results of TCAR are encouraging, they involved only 114 patients in the pivotal trial, such that further evaluation is clearly important.

There is also a body of evidence for TCAR from the SVS VQI, which demonstrates a comparable benefit/risk profile to CEA in patients in both high and standard surgical risk patients. Furthermore, TCAR has shown significantly reduced odds of certain procedural complications such as cranial nerve injury when compared to CEA as well as significantly shorter procedural times and significantly reduced odds of hospital length of stay greater than 1 day. In a recent analysis from the SVS VQI, TCAR was shown to be non-inferior to CEA in patients at standard risk for adverse events from CEA leading to FDA approval of expanded indications to include both standard and high surgical risk patients.

Objective:

The TCAR Surveillance Project is a prospective, continuous duration, case controlled, national observational registry of consecutive patients treated with TCAR using FDA-cleared proximal embolic protection devices with flow reversal and FDA-approved carotid artery stents intended for transcarotid delivery in hospitals participating in the CAS Registry of the SVS PSO VQI. This registry will provide a platform for data collection and analysis to provide ongoing surveillance of all existing and future TCAR devices.

TCAR outcomes will be compared to those of CEA in the standard and high surgical risk population as recorded in the SVS PSO VQI CEA Registry. Acute, periprocedural and long-term outcomes will be analyzed in propensity matched, risk adjusted cohorts. Standardized data elements available in both the CAS and CEA registries will be employed to make the comparisons. Participating hospitals are responsible for data entry using a secure, web-based data entry interface. Completeness and accuracy of data entry will be monitored by the SVS PSO.

The primary endpoint for both TCAR and CEA is death and/or ipsilateral carotid territory stroke at one year. The secondary endpoint will be any stroke during the initial hospitalization and death at 30 days post procedure.

Methods:

All patients, both high surgical risk and standard surgical risk patients, treated with TCAR and CEA in the SVS PSO CAS and CEA Registries will be included and separately analyzed as symptomatic and asymptomatic, with symptomatic defined as a history of ipsilateral stroke, TIA and/or amaurosis fugax within 180 days of the procedure. 30-day and one-year outcomes will be analyzed in propensity matched, risk adjusted cohorts. Any FDA-cleared proximal embolic protection device and FDA-approved carotid artery stent system indicated for the transcarotid approach will be included in the registry. Sites participating in VQI are audited for consecutive case submission by comparison with claims data. A Steering Committee within the SVS PSO will monitor the quality and completeness of submitted data, and adjudicate any questionable outcomes by querying sites for clarifying information. This committee will be responsible for scientific analysis and periodic publication of the results.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing TCAR or CEA both standard surgical risk and high surgical risk as defined by the CMS criteria published in the National Coverage Determination for Percutaneous Transluminal Angioplasty (20.7).

Exclusion Criteria:

* Patients who have received a previous stent in the target artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo TCAR and CEA in hospitals participating in the CAS or CEA registries of the SVS PSO
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year ipsilateral stroke or death | 1 year
  Any death or stroke in the territory of the treated carotid artery within one year of the carotid artery treatment

SECONDARY OUTCOMES:
30-day Stroke or death | 30 days
  Any stroke or death within 30 days of the carotid artery treatment
30-day Stroke, death or myocardial infarction | 30 days
  Any stroke, death or myocardial infarction within 30 days of the carotid artery treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Schermerhorn, MD, Study Chair — Society for Vascular Surgery Patient Safety Organization
Locations (1):
- Society for Vascular Surgery Patient Safety Organization, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schermerhorn ML, Fokkema M, Goodney P, Dillavou ED, Jim J, Kenwood CT, Siami FS, White RA; SVS Outcomes Committee. The impact of Centers for Medicare and Medicaid Services high-risk criteria on outcome after carotid endarterectomy and carotid artery stenting in the SVS Vascular Registry. J Vasc Surg. 2013 May;57(5):1318-24. doi: 10.1016/j.jvs.2012.10.107. Epub 2013 Feb 11. PMID 23406712
- [Background] Kwolek CJ, Jaff MR, Leal JI, Hopkins LN, Shah RM, Hanover TM, Macdonald S, Cambria RP. Results of the ROADSTER multicenter trial of transcarotid stenting with dynamic flow reversal. J Vasc Surg. 2015 Nov;62(5):1227-34. doi: 10.1016/j.jvs.2015.04.460. PMID 26506270